CLINICAL TRIAL: NCT00410384
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, 76-Week Study to Evaluate the Efficacy and Safety of Belimumab (HGS1006, LymphoStat-B™), a Fully Human Monoclonal Anti-BLyS Antibody, in Subjects With Systemic Lupus Erythematosus (SLE)
Brief Title: A Study of Belimumab in Subjects With Systemic Lupus Erythematosus
Acronym: BLISS-76
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Human Genome Sciences Inc. (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HGS1006-C1056; BLISS-76; 110751 (Other: GSK)
Record Dates: First submitted 2006-12-08; First posted 2006-12-12 (Estimated); Results first posted 2011-05-05 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Antibodies; Autoimmune Diseases; Systemic Lupus Erythematosus; SLE; Belimumab; Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases | interventions — belimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Belimumab 1 mg/kg (Experimental): Belimumab 1 mg/kg
  Interventions: Drug: Belimumab 1 mg/kg
- Belimumab 10 mg/kg (Experimental): Belimumab 10 mg/kg
  Interventions: Drug: Belimumab 10 mg/kg

INTERVENTIONS:
Drug: Placebo — Placebo IV plus standard therapy; placebo administered on Days 0, 14, 28, and every 28 days thereafter through 72 weeks.
  Arms: Placebo
Drug: Belimumab 1 mg/kg — Belimumab 1 mg/kg IV plus standard therapy; belimumab 1 mg/kg administered on Days 0, 14, 28, and every 28 days thereafter through 72 weeks.
  Other Names: LymphoStat-B™; belimumab
  Arms: Belimumab 1 mg/kg
Drug: Belimumab 10 mg/kg — Belimumab 10 mg/kg IV plus standard therapy; belimumab 10 mg/kg administered on Days 0, 14, 28, and every 28 days thereafter through 72 weeks.
  Other Names: LymphoStat-B™; belimumab
  Arms: Belimumab 10 mg/kg

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, tolerability, and impact on quality of life of two different doses of belimumab administered in addition to standard therapy in subjects with active, autoantibody-positive systemic lupus erythematosus (SLE) disease.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of SLE by ACR criteria.
* Active SLE disease.
* Autoantibody-positive.
* On stable SLE treatment regimen.

Key Exclusion Criteria:

* Pregnant or nursing
* Have received treatment with any B cell targeted therapy.
* Have received treatment with a biological investigational agent in the past year.
* Have received IV cyclophosphamide within 180 days of Day 0.
* Have severe lupus kidney disease.
* Have active central nervous system (CNS) lupus.
* Have required management of acute or chronic infections within the past 60 days.
* Have current drug or alcohol abuse or dependence.
* Have a historically positive test or test positive at screening for HIV, hepatitis B, or hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 819 (Actual)
Dates: Start 2006-12; Primary Completion 2009-09 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — Human Genome Sciences Inc.
Locations (146):
- United States (67):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Arthritis and Rheumatology Research, PPLC, Paradise Valley, Arizona
  - The University of Arizona Arthritis Center, Tucson, Arizona
  - Talbert Medical Group, Huntington Beach, California
  - Valerius Medical Group & Research Ctr of Greater Long Beach, Inc., Long Beach, California
  - University of Southern California, Los Angeles, California
  - Wallace Rheumatic Study Center, Los Angeles, California
  - UCLA Rheumatology, Los Angeles, California
  - Arthritis Care Center, Inc., San Jose, California
  - Inland Rheumatic Disease Specialties, Upland, California
  - Arthritis Associates of Colorado Springs, Colorado Springs, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Arthritis and Rheumatic Disease Specialties, Aventura, Florida
  - University of Miami-Division of Rheumatology and Immunology, Miami, Florida
  - Rheumatology Associates of Central Florida, Orlando, Florida
  - Southwest Florida Clinical Research Center, Tampa, Florida
  - Tampa Medical Group, P.A., Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Selah Medical Clinical Research Unit, Boise, Idaho
  - Rheumatology Associates, SC, Chicago, Illinois
  - University of Chicago Hospitals, Chicago, Illinois
  - Medical Specialists Clinical Research, Munster, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - Kentuckiana Center for Better Bone and Joint Health, Louisville, Kentucky
  - Ochsner Clinic Foundation, Baton Rouge, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Osteoporosis and Clinical Trials Center, Cumberland, Maryland
  - Osteoporosis & Clinical Trials Center, Hagerstown, Maryland
  - Tufts - New England Medical Center, Boston, Massachusetts
  - University of Michigan Medical Center - Regents of University of Michigan, Ann Arbor, Michigan
  - Fiechtner Research, Inc., Lansing, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Stafford Medical Associates, PA, Dover, New Hampshire
  - SUNY-Downstate Medical Center, Brooklyn, New York
  - North Shore-LIJ Health System/Rheumatology and Allergy Clinic, Lake Success, New York
  - Feinstein Institute, Manhasset, New York
  - Hopital for Joint Diseases, New York, New York
  - Hospital for Special Surgery, New York, New York
  - AAIR Research Center, Rochester, New York
  - Rheumatology Associates, Smithtown, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Physicians East, PA, Greenville, North Carolina
  - Wake Forest University Health Services, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - STAT Research, Inc., Dayton, Ohio
  - Oklahoma Medical Research Center, Oklahoma City, Oklahoma
  - Oklahoma Center For Arthritis Therapy & Research, Tulsa, Oklahoma
  - East Penn Rheumatology Associates, Bethlehem, Pennsylvania
  - Altoona Center for Clinical Research, Duncanville, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Low Country Rheumatology, PA/Low Country Research Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Clinical Trial at Piedmont Arthritis Clinic, Greenville, South Carolina
  - Walter Chase, Austin, Texas
  - University of Texas - Southwestern Medical Center, Dallas, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - The Rheumatic Disease Clinical Research Center, Houston, Texas
  - Accurate Clinical Research, Houston, Texas
  - Houston Institute for Clinical Research, Houston, Texas
  - Arthritis Center of South Texas, San Antonio, Texas
  - Texas Research Center, Sugar Land, Texas
  - Rheumatology Clinic, Salt Lake City, Utah
  - Arthritis Clinic of Northern Virginia, P.C., Arlington, Virginia
  - The Seattle Arthritis Clinic, Seattle, Washington
  - Arthritis Northwest, PLLC, Spokane, Washington
  - Gundersen Clinic, Ltd., Onalaska, Wisconsin
- Austria (2):
  - Universitatsklinik fur innere Medizin, Graz
  - Rheumazentrum Favoriten, Vienna
- Belgium (3):
  - Cliniques Universitaires, Brussels
  - University Hospital, Leuven
  - CHU Sart Tilman, Liège
- Canada (3):
  - Toronto Western Hospital, Toronto, Ontario
  - Centre for Prognosis Studies in Rheaumatic Diseases, Toronto, Ontario
  - McGill University Health Centre, Montreal General Hospital, Montreal
- Hospital Clinica Biblica, San José, Costa Rica
- Czechia (4):
  - University Hospital Brno, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital Olomouc, Olomouc
  - Institute of Rheumatology, Prague
- France (5):
  - CHU Hospital de Bicetre, Le Kremlin-Bicêtre
  - Hospital Huriez, Lille
  - Nouvel Hospital Civil - Medecine Interne et Immunologie Clinique, Stasbourg
  - Hospital FOCH, Suresnes
  - Centre Hospitalier Universitarie (CHU) - PURPAA, Toulouse
- Germany (13):
  - Kerckhoff-Klink Bad Nauheim, Bad Nauheim
  - Schlossparkklinik, Berlin
  - Charite, Berlin
  - Uniklinik Dusseldorf-Klinik for Endokrinologie, Diabetologie and Rheumatologie Klinik, Düsseldorf
  - FA Universitat Erlangen Nurnberg, Erlangen
  - Universitatsklinikum Frankfurt, Frankfurt
  - Medizinische Universitatsklinik, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - Friedrich Schiller Universitat, Jena
  - Universitatsklinik Schleswig-Holstein, Campus Kiel, Kiel
  - Universitatsklinikum Leipzig, Leipzig
  - Universitatsklinik Mainz, Mainz
  - Universitatsklinikum Tubingen, Tübingen
- Israel (8):
  - Soroka University Medical Center, Beersheba
  - B'nai-Zion Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Beilinson Hospital, Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel-Aviv Saurasky Medical Center, Tel Aviv
- Italy (8):
  - A. O. Ospedaliera-Universitaria Arcispedale, Ferrara
  - A.O. Ospedale San Carlo Borromeo, Milan
  - Policlinico di Modena, Modena
  - Policlinico Universitario of Padova, Padua
  - A.O. San Camillo, Rome
  - Policlinico Umberto 1, Rome
  - U.O. di reumatologia Presidio Ospedaliero di Scafati, Scafati
  - Azienda Ospedaliero University-Santa Maria della Misericordia, Udine
- Mexico (7):
  - Hospital Civil de Guadalajara "Fray Antonio Alcalde", Guadalajara
  - Instituto Jalisciense de Investigacion Clinica, Jalisco
  - Hospital General de México, Mexico City
  - Hospital Regional 1o de Octubre - ISSSTE, Mexico City
  - Insituto Nacional de Ciencias Medicas y Nutricion Salvador Zubirin, Mexico City
  - Hospital Central de S.L.P. "Iganico Morones Prieto", San Luis Potosí City
  - Instituto de Seguridad Social del Estado de Mexico y Municipios, Toluca
- Netherlands (4):
  - Leiden University Medical Center, Leiden
  - University Medical Center Maastricht, Maastricht
  - Erasmus Medical Center, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
- Poland (6):
  - Szpital Uniwerytecki nr Zim. dr. Jana Biziela, Bydgoszcz
  - Szpital Specjalistyczny Sw. Lukasza, Gmina Końskie
  - Malopolskie Centrum Medyczne, Krakow
  - Gabinety Profesorow Osrodek Baden Klinicznych, Lublin
  - Klinika Reumatologii im Prof. Eleonory Reicher, Warsaw
  - Akademicki Szpital Klinika Reumatologii Chorob Wewnetrznych, Wroclaw
- Puerto Rico (2):
  - Ponce School of Medicine, Ponce
  - University of Puerto Rico Medical Center, Rio Piedras
- Romania (2):
  - Spitalul Clinic "Sf Maria", Bucharest
  - Spitalul Clinic Colentina, Bucharest
- Narodny Ustav Reumatickych Chorob, Piešťany, Slovakia
- Spain (6):
  - Hospital La Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial Barcelona, Barcelona
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitario La Paz, Madrid
  - Hospital Son Dureta, Mallorca
  - Hospital Regional Universitario de SAS - Carlos Haya, Málaga
- Sweden (2):
  - Sahlgrensja University Hospital, Gothenburg
  - Karolinska Universitetssjukhuset, Stockholm
- United Kingdom (2):
  - St. Thomas Hospital, London
  - Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Botto J, Cetrez N, Nikolopoulos D, Regardt M, Heintz E, Lindblom J, Parodis I. Predicting EQ-5D full health state in systemic lupus erythematosus using machine learning algorithms. Rheumatol Adv Pract. 2025 Apr 18;9(2):rkaf032. doi: 10.1093/rap/rkaf032. eCollection 2025. PMID 40256631
- [Derived] Nikolopoulos D, Cetrez N, Lindblom J, Parodis I. Neuropsychiatric involvement in systemic lupus erythematosus contributes to organ damage beyond the nervous system: a post-hoc analysis of 5 phase III randomized clinical trials. Rheumatol Int. 2024 Sep;44(9):1679-1689. doi: 10.1007/s00296-024-05667-5. Epub 2024 Aug 8. PMID 39115551
- [Derived] Arends EJ, Zlei M, Tipton CM, Cotic J, Osmani Z, de Bie FJ, Kamerling SWA, van Maurik A, Dimelow R, Gregan YI, Fox NL, Rabelink TJ, Roth DA, Sanz I, van Dongen JJM, van Kooten C, Teng YKO. Disruption of memory B-cell trafficking by belimumab in patients with systemic lupus erythematosus. Rheumatology (Oxford). 2024 Sep 1;63(9):2387-2398. doi: 10.1093/rheumatology/keae286. PMID 38775637
- [Derived] Jesus D, Henriques C, Matos A, Doria A, Ines LS. Systemic Lupus Erythematosus Disease Activity Score Remission and Low Disease Activity States Discriminate Drug From Placebo and Better Health-Related Quality of Life. Arthritis Care Res (Hoboken). 2024 Jun;76(6):788-795. doi: 10.1002/acr.25305. Epub 2024 Feb 29. PMID 38258369
- [Derived] Jagerback S, Gomez A, Parodis I. Predictors of renal flares in systemic lupus erythematosus: a post-hoc analysis of four phase III clinical trials of belimumab. Rheumatology (Oxford). 2025 Feb 1;64(2):623-631. doi: 10.1093/rheumatology/keae023. PMID 38216728
- [Derived] Gomez A, Jagerback S, Sjowall C, Parodis I. Belimumab and antimalarials combined against renal flares in patients treated for extra-renal systemic lupus erythematosus: results from 4 phase III clinical trials. Rheumatology (Oxford). 2024 Feb 1;63(2):338-348. doi: 10.1093/rheumatology/kead253. PMID 37228028
- [Derived] Emamikia S, Oon S, Gomez A, Lindblom J, Borg A, Enman Y, Morand E, Grannas D, van Vollenhoven RF, Nikpour M, Parodis I. Impact of remission and low disease activity on health-related quality of life in patients with systemic lupus erythematosus. Rheumatology (Oxford). 2022 Nov 28;61(12):4752-4762. doi: 10.1093/rheumatology/keac185. PMID 35302581
- [Derived] Gupta SV, Fanget MC, MacLauchlin C, Clausen VA, Li J, Cloutier D, Shen L, Robbie GJ, Mogalian E. Clinical and Preclinical Single-Dose Pharmacokinetics of VIR-2218, an RNAi Therapeutic Targeting HBV Infection. Drugs R D. 2021 Dec;21(4):455-465. doi: 10.1007/s40268-021-00369-w. Epub 2021 Nov 6. PMID 34741731
- [Derived] Zhou X, Lee TI, Zhu M, Ma P. Prediction of Belimumab Pharmacokinetics in Chinese Pediatric Patients with Systemic Lupus Erythematosus. Drugs R D. 2021 Dec;21(4):407-417. doi: 10.1007/s40268-021-00363-2. Epub 2021 Oct 9. PMID 34628605
- [Derived] Brunner HI, Abud-Mendoza C, Mori M, Pilkington CA, Syed R, Takei S, Viola DO, Furie RA, Navarra S, Zhang F, Bass DL, Eriksson G, Hammer AE, Ji BN, Okily M, Roth DA, Quasny H, Ruperto N. Efficacy and safety of belimumab in paediatric and adult patients with systemic lupus erythematosus: an across-study comparison. RMD Open. 2021 Sep;7(3):e001747. doi: 10.1136/rmdopen-2021-001747. PMID 34531304
- [Derived] Rendas-Baum R, Baranwal N, Joshi AV, Park J, Kosinski M. Psychometric properties of FACIT-Fatigue in systemic lupus erythematosus: a pooled analysis of three phase 3 randomised, double-blind, parallel-group controlled studies (BLISS-SC, BLISS-52, BLISS-76). J Patient Rep Outcomes. 2021 Apr 8;5(1):33. doi: 10.1186/s41687-021-00298-x. PMID 33830377
- [Derived] Maslen T, Bruce IN, D'Cruz D, Ianosev M, Bass DL, Wilkinson C, Roth DA. Efficacy of belimumab in two serologically distinct high disease activity subgroups of patients with systemic lupus erythematosus: post-hoc analysis of data from the phase III programme. Lupus Sci Med. 2021 Feb;8(1):e000459. doi: 10.1136/lupus-2020-000459. PMID 33568389
- [Derived] Gomez A, Hani Butrus F, Johansson P, Akerstrom E, Soukka S, Emamikia S, Enman Y, Pettersson S, Parodis I. Impact of overweight and obesity on patient-reported health-related quality of life in systemic lupus erythematosus. Rheumatology (Oxford). 2021 Mar 2;60(3):1260-1272. doi: 10.1093/rheumatology/keaa453. PMID 32918459
- [Derived] van Vollenhoven RF, Navarra SV, Levy RA, Thomas M, Heath A, Lustine T, Adamkovic A, Fettiplace J, Wang ML, Ji B, Roth D. Long-term safety and limited organ damage in patients with systemic lupus erythematosus treated with belimumab: a Phase III study extension. Rheumatology (Oxford). 2020 Feb 1;59(2):281-291. doi: 10.1093/rheumatology/kez279. PMID 31302695
- [Derived] Furie RA, Wallace DJ, Aranow C, Fettiplace J, Wilson B, Mistry P, Roth DA, Gordon D. Long-Term Safety and Efficacy of Belimumab in Patients With Systemic Lupus Erythematosus: A Continuation of a Seventy-Six-Week Phase III Parent Study in the United States. Arthritis Rheumatol. 2018 Jun;70(6):868-877. doi: 10.1002/art.40439. Epub 2018 Apr 25. PMID 29409143
- [Derived] Furie R, Petri MA, Strand V, Gladman DD, Zhong ZJ, Freimuth WW; BLISS-52 and BLISS-76 Study Groups. Clinical, laboratory and health-related quality of life correlates of Systemic Lupus Erythematosus Responder Index response: a post hoc analysis of the phase 3 belimumab trials. Lupus Sci Med. 2014 Jun 26;1(1):e000031. doi: 10.1136/lupus-2014-000031. eCollection 2014. PMID 25396065
- [Derived] Petri MA, van Vollenhoven RF, Buyon J, Levy RA, Navarra SV, Cervera R, Zhong ZJ, Freimuth WW; BLISS-52 and BLISS-76 Study Groups. Baseline predictors of systemic lupus erythematosus flares: data from the combined placebo groups in the phase III belimumab trials. Arthritis Rheum. 2013 Aug;65(8):2143-53. doi: 10.1002/art.37995. PMID 23754628
- [Derived] Strand V, Levy RA, Cervera R, Petri MA, Birch H, Freimuth WW, Zhong ZJ, Clarke AE; BLISS-52 and -76 Study Groups. Improvements in health-related quality of life with belimumab, a B-lymphocyte stimulator-specific inhibitor, in patients with autoantibody-positive systemic lupus erythematosus from the randomised controlled BLISS trials. Ann Rheum Dis. 2014 May;73(5):838-44. doi: 10.1136/annrheumdis-2012-202865. Epub 2013 Mar 22. PMID 23524886
- [Derived] Wallace DJ, Navarra S, Petri MA, Gallacher A, Thomas M, Furie R, Levy RA, van Vollenhoven RF, Cooper S, Zhong ZJ, Freimuth W, Cervera R; BLISS-52 and -76, and LBSL02 Study Groups. Safety profile of belimumab: pooled data from placebo-controlled phase 2 and 3 studies in patients with systemic lupus erythematosus. Lupus. 2013 Feb;22(2):144-54. doi: 10.1177/0961203312469259. Epub 2012 Dec 4. PMID 23213069
- [Derived] Chatham WW, Wallace DJ, Stohl W, Latinis KM, Manzi S, McCune WJ, Tegzova D, McKay JD, Avila-Armengol HE, Utset TO, Zhong ZJ, Hough DR, Freimuth WW, Migone TS; BLISS-76 Study Group. Effect of belimumab on vaccine antigen antibodies to influenza, pneumococcal, and tetanus vaccines in patients with systemic lupus erythematosus in the BLISS-76 trial. J Rheumatol. 2012 Aug;39(8):1632-40. doi: 10.3899/jrheum.111587. Epub 2012 Jun 15. PMID 22707609
- [Derived] van Vollenhoven RF, Petri MA, Cervera R, Roth DA, Ji BN, Kleoudis CS, Zhong ZJ, Freimuth W. Belimumab in the treatment of systemic lupus erythematosus: high disease activity predictors of response. Ann Rheum Dis. 2012 Aug;71(8):1343-9. doi: 10.1136/annrheumdis-2011-200937. Epub 2012 Feb 15. PMID 22337213
- [Derived] Stohl W, Hiepe F, Latinis KM, Thomas M, Scheinberg MA, Clarke A, Aranow C, Wellborne FR, Abud-Mendoza C, Hough DR, Pineda L, Migone TS, Zhong ZJ, Freimuth WW, Chatham WW; BLISS-52 Study Group; BLISS-76 Study Group. Belimumab reduces autoantibodies, normalizes low complement levels, and reduces select B cell populations in patients with systemic lupus erythematosus. Arthritis Rheum. 2012 Jul;64(7):2328-37. doi: 10.1002/art.34400. PMID 22275291
- [Derived] Furie R, Petri M, Zamani O, Cervera R, Wallace DJ, Tegzova D, Sanchez-Guerrero J, Schwarting A, Merrill JT, Chatham WW, Stohl W, Ginzler EM, Hough DR, Zhong ZJ, Freimuth W, van Vollenhoven RF; BLISS-76 Study Group. A phase III, randomized, placebo-controlled study of belimumab, a monoclonal antibody that inhibits B lymphocyte stimulator, in patients with systemic lupus erythematosus. Arthritis Rheum. 2011 Dec;63(12):3918-30. doi: 10.1002/art.30613. PMID 22127708
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: HGS1006-C1056 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: HGS1006-C1056 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: HGS1006-C1056 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: HGS1006-C1056 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: HGS1006-C1056 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: HGS1006-C1056 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: HGS1006-C1056 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Belimumab 1 mg/kg | Belimumab 10 mg/kg
Started | 275 | 271 | 273
Completed | 186 | 199 | 191
Not Completed | 89 | 72 | 82
Not completed — Withdrawal by Subject | 28 | 17 | 20
Not completed — Adverse Event | 23 | 18 | 23
Not completed — Lack of Efficacy | 20 | 12 | 17
Not completed — Lack of Compliance | 2 | 2 | 2
Not completed — Lost to Follow-up | 4 | 6 | 6
Not completed — Protocol Violation | 6 | 6 | 6
Not completed — Physician Decision | 3 | 3 | 4
Not completed — Other | 3 | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Belimumab 1 mg/kg | Belimumab 10 mg/kg | Total
Number analyzed (Participants) | 275 | 271 | 273 | 819
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (11.9) | 40.0 (11.4) | 40.5 (11.1) | 40.2 (11.5)
Age, Customized [Number; unit: participants]
  ≤ 45 years | 189 | 184 | 178 | 551
  Between 45 and 65 years | 77 | 83 | 92 | 252
  ≥ 65 years | 9 | 4 | 3 | 16
Gender [Count of Participants; unit: Participants]
  Female | 252 | 253 | 259 | 764
  Male | 23 | 18 | 14 | 55
Region of Enrollment [Number; unit: participants]
  North America | 145 | 155 | 136 | 436
  Europe | 100 | 90 | 105 | 295
  Central America | 30 | 26 | 32 | 88

OUTCOME MEASURES:

1. Primary Outcome: SLE Responder Index (SRI) Response Rate at Week 52
Description: Percentage of subjects with a ≥ 4 point reduction from baseline in SELENA SLEDAI score, and no worsening (increase of < 0.30 points from baseline) in PGA, and no new BILAG A organ domain score or 2 new BILAG B organ domain scores compared with baseline.
  SELENA SLEDAI is calculated from 24 individual descriptors; 0 indicates inactive disease and the maximum theoretical score is 105; scores > 20 are rare. PGA is a visual analog scale scored from 0 to 3 (1=mild, 2=moderate, 3=severe). BILAG uses a single score for each of the 8 organ domains; range is from severe to no disease (A to E).
Time Frame: Baseline, 52 Weeks
Population: Analysis was performed on a modified intention-to-treat (MITT) population, defined as all subjects who were randomized and received at least 1 dose of study agent. Subjects who required rescue SLE medications were declared nonresponders, as were subjects who dropped out or were missing Week 52 data.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Belimumab 1 mg/kg | Belimumab 10 mg/kg
Number analyzed (Participants) | 275 | 271 | 273
Percentage of participants | 33.5 | 40.6 | 43.2
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Superiority or Other; p = 0.0167, Regression, Logistic — For the primary analysis of the primary efficacy endpoint, a step-down sequential testing procedure was used to control the type 1 error; Adjusted for baseline stratification factors (SELENA SLEDAI Score: ≤9 vs ≥10; proteinuria: <2g vs ≥2g per 24hr; Race: African/indig-American vs Other); Odds Ratio (OR) = 1.54, 95% CI 2-sided [1.08 to 2.19]
Statistical Analysis 2: Comparison: Placebo vs Belimumab 1 mg/kg; Test type: Superiority or Other; p = 0.0889, Regression, Logistic — After superiority of 10 mg/kg vs placebo was established, the 1 mg/kg group was tested vs placebo (2-sided alpha=0.05); Adjusted for baseline stratification factors; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.95 to 1.94]

2. Secondary Outcome: SRI Response Rate at Week 76
Description: as for outcome 1
Time Frame: Baseline, 76 Weeks
Population: Analysis was performed on a MITT population, defined as all subjects who were randomized and received at least 1 dose of study agent. Subjects who required rescue SLE medications were declared nonresponders, as were subjects who dropped out or were missing Week 76 data.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Belimumab 1 mg/kg | Belimumab 10 mg/kg
Number analyzed (Participants) | 275 | 271 | 273
Percentage of participants | 32.4 | 39.1 | 38.5
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Superiority or Other; p = 0.1323, Regression, Logistic; Analysis was adjusted for baseline stratification factors; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.92 to 1.87]
Statistical Analysis 2: Comparison: Placebo vs Belimumab 1 mg/kg; Test type: Superiority or Other; p = 0.1050, Regression, Logistic; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.94 to 1.91] — Analysis was adjusted for baseline stratification factors

3. Secondary Outcome: Percent of Subjects With a ≥ 4 Point Reduction From Baseline in SELENA SLEDAI Score at Week 52.
Time Frame: Baseline, 52 Weeks
Population: Analysis was performed on a MITT population, defined as all subjects who were randomized and received at least 1 dose of study agent.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Belimumab 1 mg/kg | Belimumab 10 mg/kg
Number analyzed (Participants) | 275 | 271 | 273
Percentage of participants | 35.3 | 42.8 | 46.5
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Superiority or Other; p = 0.0063, Regression, Logistic; Adjusted for baseline stratification factors; Odds Ratio (OR) = 1.63, 95% CI 2-sided [1.15 to 2.32]
Statistical Analysis 2: Comparison: Placebo vs Belimumab 1 mg/kg; Test type: Superiority or Other; p = 0.0740, Regression, Logistic; Adjusted for baseline stratification factors; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.97 to 1.96]

4. Secondary Outcome: Mean Change in Physician's Global Assessment (PGA) at Week 24.
Description: The PGA is a visual analog scale scored from 0 to 3. A score of 1 corresponds to mild lupus disease activity. A score of 2 correlates with moderate disease activity and a score of 3 with severe disease activity.
Time Frame: Baseline, 24 Weeks
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Scores on a 3-point scale
Arm/Group | Placebo | Belimumab 1 mg/kg | Belimumab 10 mg/kg
Number analyzed (Participants) | 275 | 271 | 273
Scores on a 3-point scale | -0.49 (0.04) | -0.47 (0.04) | -0.44 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Superiority or Other; p = 0.7962, ANCOVA; Adjusted for baseline PGA and baseline stratification factors
Statistical Analysis 2: Comparison: Placebo vs Belimumab 1 mg/kg; Test type: Superiority or Other; p = 0.9703, ANCOVA; Adjusted for baseline PGA and baseline stratification factors

5. Secondary Outcome: Mean Change From Baseline in Medical Outcomes 36-Item Short Form Health Survey (SF-36) Physical Component Summary Score (PCS) at Week 24.
Description: The SF-36 is a generic health related quality of life (HRQOL) measurement. The survey includes 36 questions grouped to 8 domains and 2 summary measures (physical and mental health component, PCS and MCS, respectively) assessing HRQOL. Responses are scored according to the SF-36v2™ manual. A score is calculated for each SF-36 domain based on the patient's response to each question within it. This is then transformed to a scale ranging from 0 (worst) to 100 (best) points. The PCS is norm-based where the mean=50 and standard deviation (SD)=10. Higher scores represent better physical health.
Time Frame: Baseline, 24 Weeks
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Belimumab 1 mg/kg | Belimumab 10 mg/kg
Number analyzed (Participants) | 275 | 271 | 273
Scores on a scale | 3.35 (0.51) | 3.78 (0.46) | 3.21 (0.43)
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Superiority or Other; p = 0.6583, ANCOVA; Analysis adjusted for baseline PCS and baseline stratification factors
Statistical Analysis 2: Comparison: Placebo vs Belimumab 1 mg/kg; Test type: Superiority or Other; p = 0.3762, ANCOVA; Analysis adjusted for baseline PCS and baseline stratification factors

6. Secondary Outcome: Percent of Subjects Whose Average Prednisone Dose Has Been Reduced by ≥ 25% From Baseline to ≤ 7.5 mg/Day During Weeks 40 Through 52
Time Frame: Baseline, Weeks 40-52
Population: Analysis was performed on a MITT population, defined as all subjects who were randomized and received at least 1 dose of study agent. Includes only subjects with baseline prednisone dose > 7.5 mg/day.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Belimumab 1 mg/kg | Belimumab 10 mg/kg
Number analyzed (Participants) | 126 | 130 | 120
Percentage of participants | 12.7 [lower limit 0.78] | 19.2 | 17.5
Statistical Analysis 1: Comparison: Placebo vs Belimumab 10 mg/kg; Test type: Superiority or Other; p = 0.4253, Regression, Logistic; Analysis was adjusted for baseline prednisone dose and baseline stratification factors; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.65 to 2.74]
Statistical Analysis 2: Comparison: Placebo vs Belimumab 1 mg/kg; Test type: Superiority or Other; p = 0.2081, Regression, Logistic; Analysis was adjusted for baseline prednisone dose and baseline stratification factors; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.78 to 3.13]

7. Other Pre Specified Outcome: Adverse Event (AE) Overview
Description: SEE ALSO ADVERSE EVENT RESULTS SECTION
Time Frame: Up to 80 Weeks
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Belimumab 1 mg/kg | Belimumab 10 mg/kg
Number analyzed (Participants) | 275 | 271 | 273
Percentage of participants
  Percent of patients with at least 1 AE | 92.0 | 93.4 | 92.7
  Percent of patients with at least 1 Serious AE | 19.6 | 23.2 | 22.3
  Percent of patients with an AE resulting in death | 0.0 | 0.7 | 0.4

ADVERSE EVENTS:
Time Frame: Up to 80 weeks
Description: Includes AEs reported in patients from first dose of study agent throughout the study up to the Week 76/Exit visit or 8 weeks following the last dose of study agent for patients who withdrew from this study or decided not to participate in the optional continuation protocol (HGS1006-C1066/NCT00724867 or HGS 1006-C1074/NCT00712933).
Arm/Group | Placebo | Belimumab 1 mg/kg | Belimumab 10 mg/kg
Serious Adverse Events (participants affected / at risk) | 54/275 | 63/271 | 61/273
Other Adverse Events (participants affected / at risk) | 213/275 | 217/271 | 219/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=275) | Belimumab 1 mg/kg (N=271) | Belimumab 10 mg/kg (N=273)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 1
Thymus enlargement (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Pericarditis lupus (Cardiac disorders) | 0 | 1 | 0
Prinzmetal angina (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Chorioretinopathy (Eye disorders) | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Chest discomfort (General disorders) | 1 | 0 | 1
Chills (General disorders) | 0 | 1 | 0
Death (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 0
Infusion related reaction (General disorders) | 0 | 1 | 3
Non-cardiac chest pain (General disorders) | 4 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 2
Pyrexia (General disorders) | 2 | 1 | 4
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 3 | 2 | 1
Gallbladder non-functioning (Hepatobiliary disorders) | 0 | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 3
Bronchitis bacterial (Infections and infestations) | 0 | 1 | 0
Bursitis infective staphylococcal (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 0 | 0
Disseminated cytomegaloviral infection (Infections and infestations) | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 2 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 2 | 0
Genital herpes (Infections and infestations) | 0 | 0 | 1
Helicobacter gastritis (Infections and infestations) | 1 | 0 | 0
Hepatitis B (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 1
Herpes zoster multi-dermatomal (Infections and infestations) | 1 | 0 | 0
HIV infection (Infections and infestations) | 1 | 0 | 0
Infected bites (Infections and infestations) | 0 | 1 | 0
Infected sebaceous cyst (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Meningitis aseptic (Infections and infestations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 3 | 5
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 2 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 3 | 3
Urosepsis (Infections and infestations) | 0 | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Narcotic intoxication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 2
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Bacteria blood identified (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
SLE arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Benign soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Carcinoid tumour of the stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1
Brain stem ischaemia (Nervous system disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Intracranial hypotension (Nervous system disorders) | 0 | 0 | 1
Lupus encephalitis (Nervous system disorders) | 1 | 0 | 1
Mononeuropathy multiplex (Nervous system disorders) | 0 | 1 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 1
Myelitis transverse (Nervous system disorders) | 0 | 1 | 0
Neuritis (Nervous system disorders) | 0 | 1 | 0
Neuropsychiatric lupus (Nervous system disorders) | 0 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 | 0 | 0
Ruptured cerebral aneurysm (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Thalamic infarction (Nervous system disorders) | 0 | 0 | 1
Vasculitis cerebral (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 2 | 2
Drug abuse (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Mania (Psychiatric disorders) | 0 | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 2 | 0 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 1
Glomerulonephritis membranous (Renal and urinary disorders) | 0 | 0 | 1
Lupus nephritis (Renal and urinary disorders) | 5 | 2 | 3
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 2
Proteinuria (Renal and urinary disorders) | 1 | 0 | 2
Renal failure acute (Renal and urinary disorders) | 3 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 2 | 0
Cervix disorder (Reproductive system and breast disorders) | 0 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 2
Femoral artery embolism (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1
Raynaud's phenomenon (Vascular disorders) | 0 | 1 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=275) | Belimumab 1 mg/kg (N=271) | Belimumab 10 mg/kg (N=273)
Anaemia (Blood and lymphatic system disorders) | 17 | 7 | 7
Abdominal pain (Gastrointestinal disorders) | 15 | 17 | 18
Abdominal pain upper (Gastrointestinal disorders) | 9 | 19 | 11
Diarrhoea (Gastrointestinal disorders) | 28 | 34 | 33
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 16 | 6
Nausea (Gastrointestinal disorders) | 27 | 42 | 45
Vomiting (Gastrointestinal disorders) | 18 | 18 | 24
Fatigue (General disorders) | 24 | 26 | 21
Oedema peripheral (General disorders) | 21 | 26 | 25
Pyrexia (General disorders) | 19 | 22 | 27
Bronchitis (Infections and infestations) | 20 | 19 | 30
Gastroenteritis (Infections and infestations) | 11 | 15 | 14
Influenza (Infections and infestations) | 12 | 19 | 8
Nasopharyngitis (Infections and infestations) | 24 | 29 | 43
Oral herpes (Infections and infestations) | 8 | 15 | 11
Pharyngitis (Infections and infestations) | 14 | 16 | 16
Sinusitis (Infections and infestations) | 28 | 21 | 31
Upper respiratory tract infection (Infections and infestations) | 58 | 53 | 54
Urinary tract infection (Infections and infestations) | 41 | 50 | 41
Viral upper respiratory tract infection (Infections and infestations) | 12 | 17 | 13
Vulvovaginal mycotic infection (Infections and infestations) | 15 | 18 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 42 | 42 | 41
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 25 | 27
Myalgia (Musculoskeletal and connective tissue disorders) | 21 | 24 | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 12 | 24
SLE arthritis (Musculoskeletal and connective tissue disorders) | 14 | 7 | 9
Dizziness (Nervous system disorders) | 11 | 14 | 16
Headache (Nervous system disorders) | 38 | 56 | 43
Anxiety (Psychiatric disorders) | 10 | 16 | 6
Depression (Psychiatric disorders) | 10 | 14 | 19
Insomnia (Psychiatric disorders) | 13 | 26 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 21 | 26
Rash (Skin and subcutaneous tissue disorders) | 12 | 17 | 20
Hypertension (Vascular disorders) | 20 | 13 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.